CLINICAL TRIAL: NCT06899217
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of CIN-102 (Deudomperidone) in Adult Subjects With Idiopathic Gastroparesis.
Brief Title: A Study to Evaluate the Efficacy and Safety of CIN-102 (Deudomperidone) in Adult Subjects With Idiopathic Gastroparesis.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CinDome Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-102-124
Record Dates: First submitted 2025-02-14; First posted 2025-03-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Gastroparesis
Keywords: Gastroparesis; Idiopathic Gastroparesis; Vomiting; Early satiety; Bloating; Epigastric pain; Abdominal pain; Delayed gastric emptying; Dopamine receptor antagonist; Nausea; Post-prandial fullness; Stomach pain; Gastric statis; Dysmotility; Gastric motility
MeSH Terms: conditions — Gastroparesis; Vomiting; Abdominal Pain; Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CIN-102: 15mg (Experimental): 15 mg CIN-102, taken orally BID for 12 weeks
  Interventions: Drug: CIN-102 Dose 15mg
- CIN-102: 10mg (Experimental): 10 mg CIN-102, taken orally BID for 12 weeks
  Interventions: Drug: CIN-102 Dose 10mg
- Placebo for CIN-102 (Placebo Comparator): Placebo for CIN-102, taken orally BID for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-102 Dose 15mg — Twice daily for 12 weeks
  Arms: CIN-102: 15mg
Drug: Placebo — Twice daily for 12 weeks
  Arms: Placebo for CIN-102
Drug: CIN-102 Dose 10mg — Twice daily for 12 weeks
  Arms: CIN-102: 10mg

SUMMARY:
The goal of this clinical trial is to evaluate if the study drug CIN-102 (deudomperidone) can help to decrease nausea severity associated with idiopathic gastroparesis severity in adult subjects.

The main questions it aims to answer are:

* To evaluate the efficacy of CIN-102 on symptoms of gastroparesis when given to patients with idiopathic gastroparesis compared to a placebo
* To evaluate the safety of CIN-102 when given to patients with idiopathic gastroparesis compared to a placebo

Participants will go through the following schedule:

* Pre-screening (1 visit)
* Screening & Lead-In (1-2 visits)

  * Will complete a Gastric Emptying Breath Test (GEBT)
  * Will complete daily diary and other Patient Reported Outcomes (PROs) as described in the protocol to assess eligibility for continued study participation.
* Lead-In Period (1 visit)
* 12-week treatment period (7 visits)

  * Study drug taken twice daily by mouth
  * Will complete daily diaries and other PROs as described in protocol
* 1 week follow-up (1 visit)

Researchers will compare the effects of the following treatments:

* 15 mg CIN-102, taken orally BID for 12 weeks
* 10 mg CIN-102, taken orally BID for 12 weeks
* Placebo for CIN-102, taken orally BID for 12 weeks

ELIGIBILITY:
Key Inclusion Criteria:

* Is a male or female ≥18 years of age;
* Has a current diagnosis of gastroparesis defined by the following:

  1. Persistent gastrointestinal (GI) symptoms that, in the opinion of the Investigator, are consistent with gastroparesis within 6 months prior to Screening; and
  2. Documented delayed gastric emptying as determined by gastric emptying breath test (GEBT) at Visit 2.
* Body mass index between 17 and 49 kg/m2, inclusive;
* If receiving treatment with a Food and Drug Administration (FDA)-approved and marketed glucagon-like peptide-1 receptor agonist (GLP-1RA) for weight loss or reduce risk of major adverse cardiovascular events, and/or, receiving any other agent(s) taken for weight loss, subjects may be considered for the study if ALL of the following criteria are satisfied:

  1. Is not taking the agent(s) for the management of diabetes or blood glucose;
  2. Has been on a stable dose of the agent(s) for at least 3 months before Screening and is expected to maintain the same dose throughout the study, including during GEBT;
  3. Is tolerating the agent(s) well, according to the Investigator's judgment;
  4. In the opinion of the Investigator, the study-qualifying signs/symptoms of gastroparesis are NOT solely due to the the agent(s); and
  5. Symptoms of gastroparesis were present before starting the agent(s).

     -------------------------------------------------------------------------

     Key Exclusion Criteria:
* Has a known primary cause of gastroparesis (eg, diabetes, surgery; acute, ongoing, or active viral illness; cancer, medications, musculoskeletal or connective tissue disorders [eg, scleroderma, systemic lupus erythematosus], or other neurologic disorder [eg, Parkinson's disease], postural orthostatic tachycardia syndrome (POTS), etc.]);
* Has a current diagnosis of Type 1 or Type 2 diabetes, according to the American Diabetes Association. Pre-diabetes is not exclusionary;
* Has been hospitalized for gastroparesis or malnutrition within 3 months prior to Screening;
* Has a known or suspected GI mechanical obstruction (eg, peptic stricture) as documented by upper GI endoscopy, upper GI radiographic series, plain film abdomen X-ray, or computed tomography (CT) in the past 2 years prior to Randomization;
* Has a history of pyloric injection of botulinum toxin within 6 months of Screening or planned injection(s) during the study;
* Has any history of pyloroplasty, pyloromyotomy, or gastric peroral endoscopic myotomy (G-POEM) procedure;
* Has a history of gastric surgery;
* Has a history of or current diagnosis of intestinal malabsorption, recurrent or chronic pancreatitis, or other pancreatic exocrine disease;
* Has a history of severe and refractory constipation;
* Has a history or evidence of clinically significant arrhythmia;
* Currently receiving parenteral feeding or presence of a nasogastric or other gastric enteral tube (e.g. percutaneous endoscopic gastrostomy [PEG] or percutaneous endoscopic jejunostomy [PEJ] tube) for feeding or decompression; Note: patients receiving enteral feeding via a jejunostomy tube may be included if, in the opinion of the Investigator, the patient is also taking substantial oral solid intake and are not primarily dependent on enteral nutrition
* Has a substance use disorder or a positive alcohol or positive drug screen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
The effect of CIN-102 to significantly decrease nausea severity as compared to baseline based on the average ANMS GCSI-DD Nausea Subscale Score. | Over the last 2 weeks of the 12-week Treatment Period as compared to Baseline
  The American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary (ANMS GCSI-DD) Nausea Subscale Scores will be averaged into a single value that ranges 0-4 (0 for no symptom and 4 for very severe).

SECONDARY OUTCOMES:
The effect of CIN-102 to significantly decrease the severity of gastroparesis-related symptoms as compared to baseline | Over the last 2 weeks of the 12-week Treatment Period as compared to Baseline
  Based on the average ANMS GCSI-DD Total Score, Composite of the Nausea and Vomiting Scores, Vomiting Score, Early Satiety Score, Postprandial Fullness Score, upper Abdominal Pain Score, and Vomiting Severity Score
The percentage of subjects who are identified as responders, defined as archiving an average ≥1 point reduction from baseline on each of ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, and individual subscale scores | Over the last 2 weeks of the 12-week Treatment Period as well as over the entire Treatment Period
  • The percentage of subjects achieving an average ≥1 point reduction from baseline, assessed separately for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, and individual subscale scores
The percentage of subjects who are identified as responders, defined as archiving an average ≥0.5 point reduction from baseline on each of ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, and individual subscale scores | Over the last 2 weeks of the 12-week Treatment Period as well as over the entire Treatment Period
  • The percentage of subjects achieving an average ≥0.5 point reduction from baseline, assessed separately for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, and individual subscale scores
The percentage of subjects who are identified as responders, defined as achieving an average ≥30% reduction from baseline for each of following: ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores | Over the last 2 weeks of the 12-week Treatment Period as well as over the entire Treatment Period
  • Occurrence of subjects achieving an average ≥ 30% reduction from baseline, assessed separately for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, and individual subscale scores
The percentage of symptom-free days in the ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores. | Over the 12-week Treatment Period
  A symptom-free day is defined as a day with severity of symptoms assessed as "none" [ie, ANMS GCSI-DD scores of 0])
The percentage of symptomatic weeks for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores | Over the 12-week Treatment Period
  A symptomatic week is defined as average ANMS GCSI-DD score ≥ 1
The percentage of mild, moderate, severe and very severe symptomatic weeks for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores | Over the 12-week Treatment Period
  Sponsor to provide definition of each severity score
The Patient Global Impression of Change (PGIC) value | Over the 12-week Treatment Period
  • The absolute change in PGIC over the 12-week Treatment Period
The Patient Global Impression of Severity (PGIS) value | From baseline to Week 12
  • The absolute change from baseline to Week 12 in PGIS
The effect of CIN-102 to significantly decrease nausea severity as compared to baseline based on the average ANMS GCSI-DD Nausea Subscale Score. | Over the final 6 weeks of the 12-week Treatment Period as compared to Baseline
  The American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary (ANMS GCSI-DD) Nausea Subscale Scores will be averaged into a single value that ranges 0-4 (0 for no symptom and 4 for very severe).
The effect of CIN-102 to significantly decrease the severity of gastroparesis-related symptoms as compared to baseline | Over the final 6 weeks of the 12-week Treatment Period as compared to Baseline
  Based on the average ANMS GCSI-DD Total Score, Composite of the Nausea and Vomiting Scores, Vomiting Score, Early Satiety Score, Postprandial Fullness Score, upper Abdominal Pain Score, and vomiting severity scores
The percentage of subjects identified as responders, defined as an average ≥0.5 reduction from baseline on each of ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores, vomiting severity scores | Over the last 6 weeks of the 12-week Treatment Period
  • Occurrence of subjects with an average ≥ 0.5 reduction from baseline, assessed separately for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores
The percentage of subjects identified as responders, defined as achieving ≥30% reduction from baseline for each: ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores, vomiting severity scores | Over the final 6 weeks of the 12-week Treatment Period
  • Occurrence of subjects achieving a ≥ 30% reduction from baseline, assessed separately for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores
The percentage of symptom-free days in the ANMS GCSI-DD Nausea Score, Total Score, Composite of the Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores | Over the final 6 weeks of the 12-week Treatment Period
  A symptom-free day is defined as a day with severity of symptoms assessed as "none" [ie, ANMS GCSI-DD scores of 0])
The percentage of symptomatic weeks for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores | Over the final 6 weeks of the 12-week Treatment Period
  A symptomatic week is defined as average ANMS GCSI-DD score ≥ 1
The percentage of moderate, severe and very severe symptomatic weeks for each of the following: ANMS GCSI-DD Nausea Score, Total Score, Composite of Nausea and Vomiting Scores, individual subscale scores, and vomiting severity scores | Over the final 6 weeks of the 12-week Treatment Period
  Sponsor to provide definition of each severity score
The Patient Global Impression of Change (PGIC) value | Over the final 6 weeks of the 12-week Treatment Period
  • The absolute change in PGIC over the 12-week Treatment Period
The Patient Global Impression of Severity (PGIS) value | Over the final 6 weeks of the 12-week Treatment Period
  • The absolute change from baseline to Week 12 in PGIS
To assess the safety of CIN-102 compared to placebo in adult subjects with idiopathic gastroparesis from the time of informed consent until the EOS | Over the 12-week Treatment Period
  * Incidence of clinically significant changes in laboratory parameters, physical examination findings, 12-lead ECG parameters, weight measurements, and vital signs, as assessed by the Investigator
  * TESAEs
  * TEAEs leading to premature discontinuation of study drug
  * Treatment-emergent clinically significant laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (85):
- United States (85):
  - Gastro Health - Birmingham, Birmingham, Alabama
  - G & L Research, LLC, Foley, Alabama
  - The Center for Clinical Trials, Saraland, Alabama
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Applied Research Center of Arkansas, Inc, Little Rock, Arkansas
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Hope Clinical Research LLC, Canoga Park, California
  - Erick H. Alayo Medical Corporation, Chula Vista, California
  - Flourish Research - Los Angeles (Covina), Covina, California
  - Gastro Care Institute, Lancaster, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - Acclaim Clinical Research, San Diego, California
  - Focus Clinical Research - West Hills, West Hills, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Rocky Mountain Gastroenterology (RMG), Lakewood, Colorado
  - Paradigm Research - Wheatridge, Wheat Ridge, Colorado
  - Connecticut Clinical Research Institute, LLC, Bristol, Connecticut
  - American Family Research Group, Cape Coral, Florida
  - USA and International Research Inc., Doral, Florida
  - Unique Clinical Trials, Doral, Florida
  - Advanced Medical Research Group, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - ENCORE Borland Groover Clinical Research, Jacksonville, Florida
  - Allied Biomedical Research Institute, Inc., Miami, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - GCP Research, St. Petersburg, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - DelRicht Clinical Research - Atlanta, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - GI Alliance - Gurnee, Gurnee, Illinois
  - Carle Clinic - Urbana Main, Urbana, Illinois
  - Integrated Clinical Trial Services, Inc, West Des Moines, Iowa
  - Kansas Medical Clinic, P.A., Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Delta Research Partners of West Monroe, LLC, Monroe, Louisiana
  - NOLA Research Works, New Orleans, Louisiana
  - Portland Gastroenterology Associates, Portland, Maine
  - Capital Digestive Care - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Sanmora Bespoke: Parkway Medical Association, Glen Burnie, Maryland
  - Gastro Health - Framingham, Framingham, Massachusetts
  - Aa Mrc, Llc, Flint, Michigan
  - Huron Gastroenterology, Ypsilanti, Michigan
  - Gastrointestinal Associates and Endoscopy Center, PA - Flowood, Flowood, Mississippi
  - KAD Clinical Research, LLC, St Louis, Missouri
  - St. Charles Clinical Research, Weldon Spring, Missouri
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Advanced Research Institute - Reno, Reno, Nevada
  - Southwest Gastroenterology Associates, Albuquerque, New Mexico
  - NY Scientific, Brooklyn, New York
  - Westchester Putnam Gastro, Carmel, New York
  - Atrium Health - Center for Gastroenterology and Hepatology MMP, Charlotte, North Carolina
  - Cross Creek Medical Clinic, PA, Fayetteville, North Carolina
  - Carolina Digestive Diseases & Endoscopy Center, Greenville, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Hometown Urgent Care and Research (Cincinnati), Cincinnati, Ohio
  - Urgent Care Specialists, LLC DBA Hometown Urgent Care and Occupational Health - Columbus, Columbus, Ohio
  - Hometown Urgent Care and Research - Huber Heights, Huber Heights, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, LLC, Westlake, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Advanced Research Institute - Portland, Portland, Oregon
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC - Smithfield, Smithfield, Pennsylvania
  - PPCP Division of Gastroenterology, Summerville, South Carolina
  - Galen Medical Group, Hixson, Tennessee
  - Digestive Health - UT Health Austin, Austin, Texas
  - Zenos Clinical Research, Dallas, Texas
  - EPIC Medical Research, DeSoto, Texas
  - Amir A Hassan, MD, PA, Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - North Hills Medical Research Inc. (North Hills Family Medicine), North Richland Hills, Texas
  - Bandera Family HealthCare Research, LLC (BFHC), San Antonio, Texas
  - GI Alliance - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Texas Digestive Specialists, Texas City, Texas
  - Advanced Research Institute - Ogden, Ogden, Utah
  - Advanced Research Institute - Sandy, Sandy City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Capital Digestive Center, Norfolk, Virginia
  - Advocate Aurora Health Research Institute, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No